CLINICAL TRIAL: NCT05505227
Title: Developing a Tailored Stigma Reduction Intervention to Increase Buprenorphine Prescribing Among Rural Primary Care Providers in Ohio
Brief Title: Developing a Tailored Stigma Reduction Intervention to Increase Buprenorphine Prescribing
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio University (Other)
Collaborators: Ohio State University (Other); Rutgers University (Other); University of North Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1R34DA057160 (NIH)
Record Dates: First submitted 2022-08-12; First posted 2022-08-17 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-04

CONDITIONS: Opioid-Related Disorders; Buprenorphine; Social Stigma; Rural Health Services
MeSH Terms: conditions — Opioid-Related Disorders; Social Stigma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Active Comparator)
  Interventions: Behavioral: Stigma-reduction training
- Control (Placebo Comparator)
  Interventions: Behavioral: Placebo

INTERVENTIONS:
Behavioral: Stigma-reduction training — While the details will be finalized by the intervention working group after the key modifiable features of OUD-stigma among rural HCPs are isolated in Aim 1, our intervention will include several new elements that distinguish it from existing stigma-reduction interventions. The prototype intervention includes several modules aimed at decreasing stigma, increasing knowledge about medications for OUD, and increasing willingness to prescribe buprenorphine (see Table 3) among rural HCPs currently in practice.
  Arms: Intervention
Behavioral: Placebo — HCPs affiliated with clinics in the control arm will receive no training but will be provided with a link to the SAMHSA website where prescribers can learn more about buprenorphine prescribing and apply to receive an X-waiver.
  Arms: Control

SUMMARY:
Buprenorphine is an evidence-based treatment for opioid use disorder that also has strong potential to reduce HIV transmission in people who use drugs. Rural health care professionals are eligible and critically needed to provide these medications, but stigma currently limits provider willingness to prescribe buprenorphine, especially in regions where mortality and HIV transmission secondary to opioid use are high. In this developmental trial, the investigators will adapt, refine, and test the feasibility of a prototype brief stigma-reduction training intervention aimed at increasing buprenorphine prescribing in the rural primary care setting.

DETAILED DESCRIPTION:
Rural counties, particularly in Appalachia, are battling fast-growing outbreaks of HIV and have been labeled by the CDC as vulnerable to growing transmission rates due to widespread injection drug use. One of the most promising mechanisms for reducing HIV transmission in these communities is the use of buprenorphine, which treats opioid use disorder and also reduces behaviors that increase HIV risk. Despite the potential benefit of buprenorphine, health care professionals (HCPs) in rural areas of the United States are much less likely to have received the training and federal waiver necessary to prescribe this medication. Stigma toward patients who use drugs is an accepted barrier to substance use treatment, but it also impacts health care professionals, especially rural primary care prescribers such as physicians, nurse practitioners, and physicians assistants who are on the front lines of the opioid crisis. The investigators have shown in previous studies that stigma is a primary reason why fewer rural health care professionals are willing to work with patients with OUD. Stigma and negative attitudes toward patients with OUD, fortunately, are modifiable but require training interventions that are both effective and feasible to implement in rural practice settings. Previous interventions have been used with health care professionals successfully to reduce stigma, but they have not been tailored for medications for opioid use, such as buprenorphine, or for the rural primary care setting. The study team proposes to adapt an existing brief stigma-reduction training intervention to the rural primary care setting to increase buprenorphine prescribing and implement a randomized, pilot study to assess feasibility and acceptability among rural primary care providers. Our specific aims are to: 1) Examine HCP knowledge and attitudes about OUD to understand their reluctance to prescribe MOUD and manage patients with OUD. 2) Develop a prototype narrative-based stigma reduction intervention and tailor it to the rural primary care setting using HCP feedback and 3) Assess the feasibility and acceptability of a stigma-reduction intervention in a pilot study in a diverse group of rural HCPs across 6 primary care clinics. The primary pilot trial outcomes are feasibility, acceptability, appropriateness, and adoption, measured among a cohort of HCPs who do not currently prescribe buprenorphine at full capacity. The investigators will also measure additional stigma outcomes such as attitudes towards patients with OUD and harm reduction. The invesstigators will use in-depth interviews to further assess perceptions of the intervention and finalize it for use in a follow-up cluster randomized controlled trial. This developmental trial will produce a brief stigma reduction training intervention that is acceptable and feasible to implement in rural primary care clinics. The long-term goal is to establish a brief stigma-reduction training intervention that is modifiable for different practice settings and effective at increasing buprenorphine prescribing in underserved communities.

ELIGIBILITY:
Inclusion Criteria:

* physician, nurse practitioner, or physician assistant
* eligible to prescribe buprenorphine under federal law
* currently practices in primary care setting
* currently practices in rural-designated county
* at least 18 years of age

Exclusion Criteria:

* currently prescribing buprenorphine at full capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility Intervention Measure | Up to 6 months
  Feasibility refers to the ease in which a new intervention can be used within a specific setting. It will be measured using the 4-item Feasibility Intervention Measure (FIM). Scale values range from 1 to 5 with higher values indicating a better outcome.
Acceptability | Up to 6 months
  Acceptability refers to HCP attitudes about whether the brief training intervention is agreeable or satisfactory. It is measured with the 4-item Acceptability of Intervention Measure (AIM) in HCP participants. Scale values range from 1 to 5 with higher values indicating a better outcome.
Appropriateness | Up to 6 months
  Appropriateness refers to the perceived alignment of the intervention within a particular practice setting and will be measured by the 4-item Intervention Appropriateness Measure (IAM). Scale values range from 1 to 5 with higher values indicating a better outcome.
Adoption | Up to 6 months
  Adoption refers to intentions or actions to adopt an EBI. Adoption will be measured as whether a HCP initiates buprenorphine prescribing for the first time or increases their patient panel (yes/no) and as the total number of patients receiving buprenorphine for each HCP.

CONTACTS AND LOCATIONS:
Overall Officials: Berkeley Franz, Ph.D., Principal Investigator — Ohio University Heritage College of Osteopathic Medicine
Locations (1):
- Berkeley Franz, Athens, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Franz B, Dhanani LY, Hall OT, Brook DL, Fenstemaker C, Simon JE, Miller WC. Buprenorphine misinformation and willingness to treat patients with opioid use disorder among primary care-aligned health care professionals. Addict Sci Clin Pract. 2024 Jan 19;19(1):7. doi: 10.1186/s13722-024-00436-y. PMID 38243307